CLINICAL TRIAL: NCT04869982
Title: A Phase IV, Randomized, Observer-blind, Placebo-controlled, Multi-center Study to Assess the Prophylactic Efficacy Against Herpes Zoster, Immunogenicity and Safety of Shingrix When Administered Intramuscularly on a 2-dose Schedule in Chinese Adults Aged 50 Years and Older
Brief Title: Efficacy, Immunogenicity and Safety Study of GSKs Recombinant Zoster Vaccine Shingrix (GSK1437173A) in Chinese Adults Aged ≥50 Years
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 212884
Record Dates: First submitted 2021-04-28; First posted 2021-05-03 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Herpes Zoster
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study was conducted in an observer-blind manner. This means that during the course of the study, the vaccine(s) recipient and those responsible for the evaluation of any study endpoint were all unaware of which study intervention was administered. The laboratory in charge of the laboratory testing was blinded to the treatment, and codes were used to link the participant and study (without any link to the treatment attributed to the participant) to each sample.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RZV Group (Experimental): Participants randomized to the RZV Group were scheduled to receive two doses of RZV, one at Day 1 and one at Month 2.
  Interventions: Biological: RZV
- Placebo Group (Placebo Comparator): Participants randomized to the Placebo Group were scheduled to receive two doses of placebo, one at Day 1 and one at Month 2.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: RZV — 2 doses of RZV in 0, 2 months schedule, administered intramuscularly in the deltoid region of the non-dominant arm
  Arms: RZV Group
Drug: Placebo — 2 doses of placebo in 0, 2 months schedule, administered intramuscularly in the deltoid region of the non-dominant arm
  Arms: Placebo Group

SUMMARY:
The purpose of this study was to assess vaccine efficacy (VE), ability to generate immune response and safety of two doses of the recombinant subunit zoster vaccine (RZV) for prevention of Herpes Zoster (HZ) in Chinese adults aged 50 years and older.

ELIGIBILITY:
Inclusion Criteria:

* Participants who, in the opinion of the investigator, can and will comply with the requirements of the protocol who, in the opinion of the investigator, can and will comply, with the requirements of the protocol.
* Written or witnessed/thumb printed informed consent obtained from the participant/participant's LAR prior to performance of any study specific procedure.
* A male or female aged 50 years or older at the time of the first vaccination.
* Medically stable participants as established by medical history and history-directed clinical examination before entering into the study.
* Female participants of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as current bilateral tubal ligation or occlusion, hysterectomy, bilateral ovariectomy or post-menopause.
* Female participants of childbearing potential may be enrolled in the study, if the subject

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series

Exclusion Criteria:

Medical conditions

* Any other condition that, in the opinion of the investigator, might interfere with the evaluations required by the study.
* History of HZ.
* Significant underlying illness that in the opinion of the investigator would be expected to prevent completion of the study
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine or study materials and equipment.
* Acute clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality as determined by physical examination or laboratory screening tests.
* Any confirmed or suspected immunosuppressive or immunodeficient condition resulting from disease or immunosuppressive/cytotoxic therapy.

Prior/Concomitant therapy

* Use of any investigational or non-registered product other than the study vaccine during the period starting 30 days before the first dose of study vaccine (Day -29 to Day 1), or planned use during the study period.
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting 30 days before each dose and ending 30 days after the last dose of vaccine administration. However, licensed pneumococcal vaccines and inactivated and subunit influenza vaccines (without adjuvant for seasonal or pandemic flu) may be co- administered with any dose of study vaccine.
* Previous vaccination against varicella or HZ.
* Administration of long-acting immune-modifying drugs at any time during the study period.
* Administration of immunoglobulins and/or any blood products or plasma derivatives during the period starting 3 months before the first dose of study vaccine up to one month post dose 2 (Month 3).
* Planned or chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting 3 months prior to the first vaccine. For corticosteroids, this will mean prednisone ≥20mg/day, or equivalent, is not allowed. Inhaled, intra-articular and topical steroids are allowed.

Prior/Concurrent clinical study experience

• Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product.

Other exclusions

* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions within 2 months of last vaccination.
* History of current/chronic alcohol consumption and/or drug abuse.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6138 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - GSK Investigational Site, Huaian, Jiangsu
  - GSK Investigational Site, Lianyungang
  - GSK Investigational Site, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD is made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf

REFERENCES:
- [Background] Alexandra Echeverria Proano D, Zhu F, Sun X, Zoco J, Soni J, Parmar N, Ali SO; Zoster-076 Study Group. Efficacy, reactogenicity, and safety of the adjuvanted recombinant zoster vaccine for the prevention of herpes zoster in Chinese adults >/= 50 years: A randomized, placebo-controlled trial. Hum Vaccin Immunother. 2024 Dec 31;20(1):2351584. doi: 10.1080/21645515.2024.2351584. Epub 2024 Jun 5. PMID 38838170
- [Derived] de Oliveira Gomes J, Gagliardi AM, Andriolo BN, Torloni MR, Andriolo RB, Puga MEDS, Canteiro Cruz E. Vaccines for preventing herpes zoster in older adults. Cochrane Database Syst Rev. 2023 Oct 2;10(10):CD008858. doi: 10.1002/14651858.CD008858.pub5. PMID 37781954

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 6 centers in China.
Pre-assignment Details: A total of 6138 participants were enrolled into the study, of which 6128 participants received at least 1 dose of study treatment/vaccine (RZV or placebo) and were included in the Exposed Set.
Period: Overall Study
Arm/Group | RZV Group | Placebo Group
Started | 3064 | 3064
Completed | 3040 | 3048
Not Completed | 24 | 16
Not completed — Consent withdrawal, not due to a (S)AE | 7 | 2
Not completed — Migrated / moved from the study area | 1 | 1
Not completed — Adverse event requiring expedited reporting | 13 | 11
Not completed — Unsolicited non-serious adverse event | 1 | 1
Not completed — Solicited adverse event | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RZV Group | Placebo Group | Total
Number analyzed (Participants) | 3064 | 3064 | 6128
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.4 (7.8) | 62.4 (7.8) | 62.4 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1868 | 1872 | 3740
  Male | 1196 | 1192 | 2388
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - East Asian Heritage | 3064 | 3064 | 6128

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Confirmed Herpes Zoster (HZ) Cases
Description: A suspected case of HZ was defined as a new unilateral rash accompanied by pain (broadly defined to include allodynia, pruritus or other sensations) and no alternative diagnosis. A confirmed case of HZ was diagnosed by Polymerase Chain Reaction (PCR) or by the HZ Ascertainment Committee (HZAC) determination. The incidence rate (n/T) of confirmed HZ cases, expressed in terms of 1000 person-years rate, was calculated as the number of participants reporting at least one confirmed HZ case (n) in a group, over the sum of follow-up period expressed in years (T) in the same group, and multiplied by 1000.
Time Frame: From Month 3 (30 days after the second vaccination) up to study end (duration of approximately 2 years)
Population: The analysis was performed on the modified Exposed Set, which excluded participants from the Exposed Set who were not administered 2 doses of the study vaccine, or who developed a confirmed case of HZ prior to 30 days after the second vaccination.
Measure: Number; unit: Cases per 1000 person-years
Arm/Group | RZV Group | Placebo Group
Number analyzed (Participants) | 2965 | 2991
Cases per 1000 person-years | 0.0 | 8.2
Statistical Analysis 1: Comparison: RZV Group vs Placebo Group; To demonstrate the vaccine efficacy (VE) of RZV against HZ, the analysis considered the exact inference on the relative risk adjusted for age strata conditionally to the total number of confirmed HZ cases observed and time at risk. This method computed an exact confidence interval (CI) around the rate ratio (ratio of the event rates in the RZV Group versus Placebo Group) and accounted for the sum of the time at risk of the participants within each group; Test type: Other — VE was defined as 1 minus the relative risk (RR). RR was defined as the ratio of the incidence rates of the RZV Group over the Placebo Group. The VE of RZV against HZ was to be demonstrated if the lower limit (LL) of the two-sided 95% CI of VE was above 25%; p < 0.0001, Poisson — All p-values reported were related to the null hypothesis test VE = 0; The CI for VE is derived from the exact CI from RR; VE (1-RR) = 100, 95% CI 2-sided [89.82 to 100]

2. Secondary Outcome: Incidence Rate of Confirmed HZ Cases, by Age Category
Description: A suspected case of HZ was defined as a new unilateral rash accompanied by pain (broadly defined to include allodynia, pruritus or other sensations) and no alternative diagnosis. A confirmed case of HZ was diagnosed by PCR or by the HZAC determination. The incidence rate (n/T) of confirmed HZ cases, expressed in terms of 1000 person-years rate, was calculated as the number of participants reporting at least one confirmed HZ case (n) in a group, over the sum of follow-up period expressed in years (T) in the same group, and multiplied by 1000. The age categories assessed were 50-69 and greater than or equal to (>=) 70 years of age (YOA).
Time Frame: From Month 3 (30 days after the second vaccination) up to study end (duration of approximately 2 years)
Population: as for outcome 1
Measure: Number; unit: Cases per 1000 person-years
Arm/Group | RZV Group | Placebo Group
Number analyzed (Participants) | 2965 | 2991
Cases per 1000 person-years
  50-69 YOA: number analyzed (Participants) | 2330 | 2360
  50-69 YOA | 0.0 | 7.4
  >=70 YOA: number analyzed (Participants) | 635 | 631
  >=70 YOA | 0.0 | 11.4

3. Secondary Outcome: Number of Participants With Any and at Least Grade 3 Solicited Local Adverse Events (AEs) (as Per GSK's Standard Grading Scale) and With Solicited Local AEs Resulting in a Medically Attended Visit
Description: Assessed solicited local AEs included erythema, pain and swelling at injection site. The intensity of a solicited local AE was scored at GSK by using GSK's standard grading scale as follows: Any AE = occurrence of the event regardless of intensity grade. At least Grade 3 AE = occurrence of an at least Grade 3 or Grade 4 event (Grade 4 defined for some solicited AEs collected in the study as required by Chinese grading scale). Maximum of Grade 3 and 4 was considered as Grade 3 for all applicable solicited symptoms in GSK standard grading table. AE resulting in a medically attended visit = event for which the participant received medical attention defined as hospitalization, or an otherwise unscheduled visit to or from medical personnel for any reason, including emergency room visits.
Time Frame: Within 7 days after each vaccination (occurring at Day 1 and Month 2)
Population: The analysis was performed on the Exposed Set, which included all participants who received at least 1 dose of the study treatment and who have documented solicited AEs after each vaccination (i.e. diary card for solicited AEs completed and returned).
Measure: Count of Participants; unit: Participants
Arm/Group | RZV Group | Placebo Group
Number analyzed (Participants) | 3053 | 3058
Participants
  Any Erythema, post-vaccination at Day 1 | 600 | 14
  At least Grade 3 Erythema, post-vaccination at Day 1 | 25 | 0
  Medically attended visit Erythema, post-vaccination at Day 1 | 8 | 0
  Any Pain, post-vaccination at Day 1 | 2045 | 217
  At least Grade 3 Pain, post-vaccination at Day 1 | 78 | 3
  Medically attended visit Pain, post-vaccination at Day 1 | 18 | 0
  Any Swelling, post-vaccination at Day 1 | 705 | 18
  At least Grade 3 Swelling, post-vaccination at Day 1 | 19 | 0
  Medically attended visit Swelling, post-vaccination at Day 1 | 11 | 0
  Any Erythema, post-vaccination at Month 2: number analyzed (Participants) | 2956 | 2987
  Any Erythema, post-vaccination at Month 2 | 375 | 9
  At least Grade 3 Erythema, post-vaccination at Month 2: number analyzed (Participants) | 2956 | 2987
  At least Grade 3 Erythema, post-vaccination at Month 2 | 7 | 0
  Medically attended visit Erythema, post-vaccination at Month 2: number analyzed (Participants) | 2956 | 2987
  Medically attended visit Erythema, post-vaccination at Month 2 | 4 | 0
  Any Pain, post-vaccination at Month 2: number analyzed (Participants) | 2956 | 2987
  Any Pain, post-vaccination at Month 2 | 1255 | 99
  At least Grade 3 Pain, post-vaccination at Month 2: number analyzed (Participants) | 2956 | 2987
  At least Grade 3 Pain, post-vaccination at Month 2 | 31 | 0
  Medically attended visit Pain, post-vaccination at Month 2: number analyzed (Participants) | 2956 | 2987
  Medically attended visit Pain, post-vaccination at Month 2 | 10 | 1
  Any Swelling, post-vaccination at Month 2: number analyzed (Participants) | 2956 | 2987
  Any Swelling, post-vaccination at Month 2 | 388 | 8
  At least Grade 3 Swelling, post-vaccination at Month 2: number analyzed (Participants) | 2956 | 2987
  At least Grade 3 Swelling, post-vaccination at Month 2 | 5 | 0
  Medically attended visit Swelling, post-vaccination at Month 2: number analyzed (Participants) | 2956 | 2987
  Medically attended visit Swelling, post-vaccination at Month 2 | 5 | 0

4. Secondary Outcome: Number of Participants With Any, at Least Grade 3 (as Per GSK's Standard Grading Scale) and Related Solicited General AEs and With Solicited General AEs Resulting in a Medically Attended Visit
Description: Assessed solicited general AEs included fatigue, fever, gastrointestinal symptoms (nausea, vomiting and/or abdominal pain) headache, myalgia, and shivering. The intensity of a solicited general AE was scored at GSK by using GSK's standard grading scale as follows: Any AE = occurrence of the event regardless of intensity grade or relation to vaccination. At least Grade 3 AE = occurrence of an at least Grade 3 or Grade 4 event (Grade 4 defined for some solicited AEs collected in the study as required by Chinese grading scale). Maximum of Grade 3 and 4 was considered as Grade 3 for all applicable solicited symptoms in GSK standard grading table. Related AE = event assessed by the investigator as related to vaccination. AE resulting in a medically attended visit = event for which the participant received medical attention defined as hospitalization, or an otherwise unscheduled visit to or from medical personnel for any reason, including emergency room visits.
Time Frame: Within 7 days after each vaccination (occurring at Day 1 and Month 2)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | RZV Group | Placebo Group
Number analyzed (Participants) | 3053 | 3058
Participants
  Any Fatigue, post-vaccination at Day 1 | 1070 | 131
  At least Grade 3 Fatigue, post-vaccination at Day 1 | 56 | 3
  Related Fatigue, post-vaccination at Day 1 | 1058 | 127
  Medically attended visit Fatigue, post-vaccination at Day 1 | 20 | 2
  Any Fever, post-vaccination at Day 1 | 260 | 14
  At least Grade 3 Fever, post-vaccination at Day 1 | 12 | 0
  Related Fever, post-vaccination at Day 1 | 259 | 14
  Medically attended visit Fever, post-vaccination at Day 1 | 10 | 3
  Any Gastrointestinal symptoms, post-vaccination at Day 1 | 331 | 51
  At least Grade 3 Gastrointestinal symptoms, post-vaccination at Day 1 | 11 | 1
  Related Gastrointestinal symptoms, post-vaccination at Day 1 | 322 | 44
  Medically attended visit Gastrointestinal symptoms, post-vaccination at Day 1 | 8 | 5
  Any Headache, post-vaccination at Day 1 | 746 | 74
  At least Grade 3 Headache, post-vaccination at Day 1 | 37 | 1
  Related Headache, post-vaccination at Day 1 | 738 | 69
  Medically attended visit Headache, post-vaccination at Day 1 | 16 | 2
  Any Myalgia, post-vaccination at Day 1 | 602 | 55
  At least Grade 3 Myalgia, post-vaccination at Day 1 | 32 | 2
  Related Myalgia, post-vaccination at Day 1 | 593 | 55
  Medically attended visit Myalgia, post-vaccination at Day 1 | 6 | 1
  Any Shivering, post-vaccination at Day 1 | 351 | 12
  At least Grade 3 Shivering, post-vaccination at Day 1 | 6 | 0
  Related Shivering, post-vaccination at Day 1 | 347 | 12
  Medically attended visit Shivering, post-vaccination at Day 1 | 7 | 1
  Any Fatigue, post-vaccination at Month 2: number analyzed (Participants) | 2956 | 2987
  Any Fatigue, post-vaccination at Month 2 | 797 | 44
  At least Grade 3 Fatigue, post-vaccination at Month 2: number analyzed (Participants) | 2956 | 2987
  At least Grade 3 Fatigue, post-vaccination at Month 2 | 32 | 0
  Related Fatigue, post-vaccination at Month 2: number analyzed (Participants) | 2956 | 2987
  Related Fatigue, post-vaccination at Month 2 | 793 | 44
  Medically attended visit Fatigue, post-vaccination at Month 2: number analyzed (Participants) | 2956 | 2987
  Medically attended visit Fatigue, post-vaccination at Month 2 | 10 | 0
  Any Fever, post-vaccination at Month 2: number analyzed (Participants) | 2956 | 2987
  Any Fever, post-vaccination at Month 2 | 284 | 6
  At least Grade 3 Fever, post-vaccination at Month 2: number analyzed (Participants) | 2956 | 2987
  At least Grade 3 Fever, post-vaccination at Month 2 | 14 | 0
  Related Fever, post-vaccination at Month 2: number analyzed (Participants) | 2956 | 2987
  Related Fever, post-vaccination at Month 2 | 283 | 6
  Medically attended visit Fever, post-vaccination at Month 2: number analyzed (Participants) | 2956 | 2987
  Medically attended visit Fever, post-vaccination at Month 2 | 7 | 1
  Any Gastrointestinal symptoms, post-vaccination at Month 2: number analyzed (Participants) | 2956 | 2987
  Any Gastrointestinal symptoms, post-vaccination at Month 2 | 190 | 20
  At least Grade 3 Gastrointestinal symptoms, post-vaccination at Month 2: number analyzed (Participants) | 2956 | 2987
  At least Grade 3 Gastrointestinal symptoms, post-vaccination at Month 2 | 1 | 1
  Related Gastrointestinal symptoms, post-vaccination at Month 2: number analyzed (Participants) | 2956 | 2987
  Related Gastrointestinal symptoms, post-vaccination at Month 2 | 186 | 19
  Medically attended visit Gastrointestinal symptoms, post-vaccination at Month 2: number analyzed (Participants) | 2956 | 2987
  Medically attended visit Gastrointestinal symptoms, post-vaccination at Month 2 | 7 | 2
  Any Headache, post-vaccination at Month 2: number analyzed (Participants) | 2956 | 2987
  Any Headache, post-vaccination at Month 2 | 575 | 26
  At least Grade 3 Headache, post-vaccination at Month 2: number analyzed (Participants) | 2956 | 2987
  At least Grade 3 Headache, post-vaccination at Month 2 | 20 | 0
  Related Headache, post-vaccination at Month 2: number analyzed (Participants) | 2956 | 2987
  Related Headache, post-vaccination at Month 2 | 573 | 26
  Medically attended visit Headache, post-vaccination at Month 2: number analyzed (Participants) | 2956 | 2987
  Medically attended visit Headache, post-vaccination at Month 2 | 10 | 2
  Any Myalgia, post-vaccination at Month 2: number analyzed (Participants) | 2956 | 2987
  Any Myalgia, post-vaccination at Month 2 | 464 | 21
  At least Grade 3 Myalgia, post-vaccination at Month 2: number analyzed (Participants) | 2956 | 2987
  At least Grade 3 Myalgia, post-vaccination at Month 2 | 20 | 0
  Related Myalgia, post-vaccination at Month 2: number analyzed (Participants) | 2956 | 2987
  Related Myalgia, post-vaccination at Month 2 | 464 | 21
  Medically attended visit Myalgia, post-vaccination at Month 2: number analyzed (Participants) | 2956 | 2987
  Medically attended visit Myalgia, post-vaccination at Month 2 | 8 | 0
  Any Shivering, post-vaccination at Month 2: number analyzed (Participants) | 2956 | 2987
  Any Shivering, post-vaccination at Month 2 | 334 | 4
  At least Grade 3 Shivering, post-vaccination at Month 2: number analyzed (Participants) | 2956 | 2987
  At least Grade 3 Shivering, post-vaccination at Month 2 | 12 | 0
  Related Shivering, post-vaccination at Month 2: number analyzed (Participants) | 2956 | 2987
  Related Shivering, post-vaccination at Month 2 | 333 | 4
  Medically attended visit Shivering, post-vaccination at Month 2: number analyzed (Participants) | 2956 | 2987
  Medically attended visit Shivering, post-vaccination at Month 2 | 5 | 0

5. Secondary Outcome: Number of Participants With at Least One Unsolicited AE, at Least One Grade 3 Unsolicited AE, at Least One Related Unsolicited AE, at Least One Grade 3 Related Unsolicited AE and With at Least One Medically Attended Unsolicited AE
Description: An unsolicited AE was defined as any AE reported in addition to those solicited during the clinical study, or any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms. At least one unsolicited AE = at least one event regardless of intensity grade or relation to study vaccination. At least one Grade 3 unsolicited AE = at least one event that prevented normal, everyday activities. At least one related unsolicited AE = at least one event assessed by the investigator as related to the study vaccination. At least one Grade 3 related unsolicited AE = at least one event that prevented normal, everyday activities assessed by the investigator as related to the study vaccination. At least one medically attended unsolicited AE = at least one event for which the participant received medical attention defined as hospitalization, or an otherwise unscheduled visit to or from medical personnel for any reason, including emergency room visits.
Time Frame: Within 30 days after any vaccination (occurring at Day 1 and Month 2)
Population: The analysis was performed on the Exposed Set, which included all participants who received at least 1 dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | RZV Group | Placebo Group
Number analyzed (Participants) | 3064 | 3064
Participants
  At least one unsolicited AE | 124 | 97
  At least one Grade 3 unsolicited AE | 8 | 10
  At least one related unsolicited AE | 31 | 17
  At least one Grade 3 related unsolicited AE | 0 | 1
  At least one medically attended unsolicited AE(s) | 64 | 53

6. Secondary Outcome: Number of Participants With at Least One Serious Adverse Event (SAE) and With at Least One Related SAE From First Vaccination (Day 1) up to 30 Days Post Last Vaccination
Description: An SAE was defined as any untoward medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity, was a congenital anomaly/birth defect in the offspring of a study participant, or resulted in abnormal pregnancy outcomes, or was considered medically significant. At least one SAE = at least one SAE regardless of relation to study vaccination. At least one related SAE = at least one SAE assessed by the investigator as related to the study vaccination.
Time Frame: From first vaccination (Day 1) up to 30 days post last vaccination (last vaccination administered at Day 1 for participants who received only 1 dose and at Month 2 for participants who received 2 doses)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RZV Group | Placebo Group
Number analyzed (Participants) | 3064 | 3064
Participants
  At least one SAE | 32 | 36
  At least one related SAE | 0 | 1

7. Secondary Outcome: Number of Participants With at Least One SAE and With at Least One Related SAE From First Vaccination (Day 1) up to 12 Months Post Last Vaccination
Description: as for outcome 6
Time Frame: From first vaccination (Day 1) up to 12 months post last vaccination (last vaccination administered at Day 1 for participants who received only 1 dose and at Month 2 for participants who received 2 doses)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RZV Group | Placebo Group
Number analyzed (Participants) | 3064 | 3064
Participants
  At least one SAE | 88 | 93
  At least one related SAE | 0 | 1

8. Secondary Outcome: Number of Participants With at Least One Related SAE From First Vaccination (Day 1) up to Study End (Duration of Approximately 2 Years)
Description: An SAE was defined as any untoward medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity, was a congenital anomaly/birth defect in the offspring of a study participant, or resulted in abnormal pregnancy outcomes, or was considered medically significant. At least one related SAE = at least one SAE assessed by the investigator as related to the study vaccination.
Time Frame: From first vaccination (Day 1) up to study end (duration of approximately 2 years)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RZV Group | Placebo Group
Number analyzed (Participants) | 3064 | 3064
Participants | 0 | 1

9. Secondary Outcome: Number of Participants With at Least One SAE Related to Study Participation or to GlaxoSmithKline Concomitant Medication/Vaccine
Description: An SAE was defined as any untoward medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity, was a congenital anomaly/birth defect in the offspring of a study participant, or resulted in abnormal pregnancy outcomes, or was considered medically significant. SAEs related to study participation (and not to the study vaccine) or to GSK concomitant medication/vaccine were assessed.
Time Frame: From the time the participant consented to participate in the study (Day 1) up to study end (duration of approximately 2 years)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RZV Group | Placebo Group
Number analyzed (Participants) | 3064 | 3064
Participants | 0 | 0

10. Secondary Outcome: Number of Participants With at Least One Fatal SAE and at Least One Related Fatal SAE From First Vaccination (Day 1) up to 30 Days Post Last Vaccination
Description: An SAE was defined as any untoward medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity, was a congenital anomaly/birth defect in the offspring of a study participant, or resulted in abnormal pregnancy outcomes, or was considered medically significant. At least one fatal SAE = at least one fatal SAE regardless of relation to study vaccination. At least one related fatal SAE = at least one fatal SAE assessed by the investigator as related to the study vaccination.
Time Frame: as for outcome 6
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RZV Group | Placebo Group
Number analyzed (Participants) | 3064 | 3064
Participants
  At least one fatal SAE | 3 | 2
  At least one related fatal SAE | 0 | 0

11. Secondary Outcome: Number of Participants With at Least One Fatal SAE and With at Least One Related Fatal SAE From First Vaccination (Day 1) up to 12 Months Post Last Vaccination
Description: as for outcome 10
Time Frame: as for outcome 7
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RZV Group | Placebo Group
Number analyzed (Participants) | 3064 | 3064
Participants
  At least one fatal SAE | 11 | 9
  At least one related fatal SAE | 0 | 0

12. Secondary Outcome: Number of Participants With at Least One Related Fatal SAE From First Vaccination (Day 1) up to Study End (Duration of Approximately 2 Years)
Description: An SAE was defined as any untoward medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity, was a congenital anomaly/birth defect in the offspring of a study participant, or resulted in abnormal pregnancy outcomes, or was considered medically significant. At least one related fatal SAE = at least one fatal SAE assessed by the investigator as related to the study vaccination.
Time Frame: From first vaccination (Day 1) up to study end (duration of approximately 2 years)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RZV Group | Placebo Group
Number analyzed (Participants) | 3064 | 3064
Participants | 0 | 0

13. Secondary Outcome: Number of Participants With at Least One Potential Immune-mediated Disease (pIMD) and at Least One Related pIMD From First Vaccination (Day 1) up to 30 Days Post Last Vaccination
Description: pIMDs were defined as a subset of AEs that included autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have had an autoimmune aetiology. At least one pIMD = at least one pIMD regardless of relation to vaccination. At least one related pIMD = at least one pIMD assessed by the investigator as related to the study vaccination.
Time Frame: as for outcome 6
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RZV Group | Placebo Group
Number analyzed (Participants) | 3064 | 3064
Participants
  At least one pIMD | 2 | 2
  At least one related pIMD | 0 | 0

14. Secondary Outcome: Number of Participants With at Least One pIMD and at Least One Related pIMD From First Vaccination (Day 1) up to 12 Months Post Last Vaccination
Description: pIMDs were defined as a subset of AEs that included autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have had an autoimmune aetiology. At least one pIMD = at least one pIMD regardless of relation to study vaccination. At least one related pIMD = at least one related pIMD assessed by the investigator as related to the study vaccination.
Time Frame: as for outcome 7
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RZV Group | Placebo Group
Number analyzed (Participants) | 3064 | 3064
Participants
  At least one pIMD | 2 | 3
  At least one related pIMD | 0 | 0

15. Secondary Outcome: Number of Participants With at Least One Related Serious pIMD From 12 Months Post Last Vaccination up to Study End (Duration of Approximately 1 Year)
Description: pIMDs were defined as a subset of AEs that included autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have had an autoimmune aetiology. At least one related serious pIMD = at least one serious pIMD assessed by the investigator as related to the study vaccination.
Time Frame: From 12 months post last vaccination (last vaccination administered at Day 1 for participants who received only 1 dose and at Month 2 for participants who received 2 doses) up to study end (duration of approximately 1 year)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RZV Group | Placebo Group
Number analyzed (Participants) | 3064 | 3064
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited local and general AEs: during the 7-day (Day 1 to Day 7) follow-up period after any vaccination; Unsolicited AEs: during the 30-day (Day 1 to Day 30) follow-up period after any vaccination; All-cause mortality and SAEs: from first vaccination (Day 1) up to study end (duration of approximately 2 years).
Description: The adverse events reported in the Other Adverse Events module were assessed based on GSK's standard grading scale.
Arm/Group | RZV Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 13/3064 | 11/3064
Serious Adverse Events (participants affected / at risk) | 90/3064 | 94/3064
Other Adverse Events (participants affected / at risk) | 2337/3064 | 485/3064
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RZV Group (N=3064) | Placebo Group (N=3064)
Agranulocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 3 (3) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 2 (2)
Arteriosclerosis coronary artery (Cardiac disorders) | 8 (9) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 1 (1)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac dysfunction (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 3 (3) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 3 (3)
Coronary artery insufficiency (Cardiac disorders) | 0 (0) | 1 (1)
Defect conduction intraventricular (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 1 (1)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Oesophageal cyst (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Thyroid mass (Endocrine disorders) | 1 (1) | 1 (1)
Thyroiditis subacute (Endocrine disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 2 (2) | 0 (0)
Diabetic blindness (Eye disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Pterygium (Eye disorders) | 2 (2) | 0 (0)
Refraction disorder (Eye disorders) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 4 (4) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 3 (3)
Peritoneal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1)
Sudden death (General disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5) | 6 (6)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Brain herniation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Craniocerebral injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Electrical burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Epidural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb crushing injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pleural injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Scapula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diabetic complication (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Lung squamous cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal ganglia haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 2 (2)
Cerebral infarction (Nervous system disorders) | 24 (24) | 18 (18)
Cerebral thrombosis (Nervous system disorders) | 0 (0) | 3 (3)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Hemiplegia (Nervous system disorders) | 1 (1) | 0 (0)
Intraventricular haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Lacunar infarction (Nervous system disorders) | 1 (1) | 1 (1)
Quadriplegia (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 2 (2) | 2 (2)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) | 1 (1)
Conversion disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 1 (1) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Urethral prolapse (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 3 (3)
Uterovaginal prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diabetic vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Essential hypertension (Vascular disorders) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 8 (9) | 4 (4)
Scalp haematoma (Vascular disorders) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 0 (0) | 2 (2)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RZV Group (N=3064) | Placebo Group (N=3064)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Porencephaly (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Deafness bilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Thyroiditis subacute (Endocrine disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastrointestinal disorder ( (Gastrointestinal disorders) | 444 (521) | 67 (71)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingival swelling (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 4 (4)
Administration site erythema (General disorders) | 762 (975) | 21 (23)
Administration site pain (General disorders) | 2203 (3300) | 280 (316)
Administration site swelling (General disorders) | 855 (1093) | 24 (26)
Axillary pain (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 2 (2) | 1 (1)
Chills (General disorders) | 544 (686) | 14 (16)
Fatigue (General disorders) | 1326 (1867) | 161 (175)
Injection site haematoma (General disorders) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 457 (544) | 21 (21)
Thirst (General disorders) | 0 (0) | 1 (1)
Vaccination site induration (General disorders) | 2 (2) | 0 (0)
Vaccination site pain (General disorders) | 1 (1) | 0 (0)
Vaccination site pruritus (General disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 9 (9) | 7 (7)
Pharyngitis (Infections and infestations) | 2 (2) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood uric acid increased (Investigations) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 811 (1067) | 71 (76)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intracranial haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular insufficiency (Nervous system disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 25 (27) | 9 (9)
Headache (Nervous system disorders) | 1001 (1321) | 94 (102)
Paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (6)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Papule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Essential hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 0 (0)
Vascular rupture (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/82/NCT04869982/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-10): https://cdn.clinicaltrials.gov/large-docs/82/NCT04869982/SAP_001.pdf